CLINICAL TRIAL: NCT02559921
Title: Safety and Immunogenicity Study of Recombinant Human Rabies Immunoglobin (rhRIG) in Combination With Rabies Vaccine for Human Use With Human Rabies Immune Globulin (HRIG) in Combination With Rabies Vaccine for Human Use in Healthy Adult Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Chaoyang District Centre for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: cycdc2015-3
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-09

CONDITIONS: Rabies
Keywords: Recombinant Human Rabies Immunoglobin (rhRIG)
MeSH Terms: conditions — Rabies | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- rhRIG（20 IU/kg）only (Experimental): Subjects received rhRIG（20 IU/kg） on day 0
  Interventions: Biological: rhRIG（20 IU/kg）
- rhRIG（40 IU/kg）only (Experimental): Subjects received rhRIG（40 IU/kg） on day 0
  Interventions: Biological: rhRIG（40 IU/kg）
- HRIG（20 IU/kg）only (Active Comparator): Subjects received HRIG（20 IU/kg）on day 0
  Interventions: Biological: HRIG（20 IU/kg）
- rhRIG（20 IU/kg）+ vaccine (Experimental): Subjects received rhRIG（20 IU/kg）in combination with rabies vaccine for human use on day 0 and received vaccine only on days 3,7,14,28
  Interventions: Biological: rhRIG（20 IU/kg） and vaccine
- rhRIG（40 IU/kg）+ vaccine (Experimental): Subjects received rhRIG（40 IU/kg）in combination with rabies vaccine for human use on day 0 and received vaccine only on days 3,7,14,28
  Interventions: Biological: rhRIG（40 IU/kg） and vaccine
- HRIG（20 IU/kg）+ vaccine (Experimental): Subjects received HRIG（20 IU/kg）in combination with rabies vaccine for human use on day 0 and received vaccine only on days 3,7,14,28
  Interventions: Biological: HRIG（20 IU/kg） and vaccine
- placebo + vaccine (Placebo Comparator): Subjects received placebo in combination with rabies vaccine for human use on day 0 and received vaccine only on days 3,7,14,28
  Interventions: Biological: placebo and vaccine

INTERVENTIONS:
Biological: rhRIG（20 IU/kg）
  Arms: rhRIG（20 IU/kg）only
Biological: rhRIG（40 IU/kg）
  Arms: rhRIG（40 IU/kg）only
Biological: HRIG（20 IU/kg）
  Arms: HRIG（20 IU/kg）only
Biological: rhRIG（20 IU/kg） and vaccine
  Arms: rhRIG（20 IU/kg）+ vaccine
Biological: rhRIG（40 IU/kg） and vaccine
  Arms: rhRIG（40 IU/kg）+ vaccine
Biological: HRIG（20 IU/kg） and vaccine
  Arms: HRIG（20 IU/kg）+ vaccine
Biological: placebo and vaccine
  Arms: placebo + vaccine

SUMMARY:
This study evaluates the rabies virus neutralizing antibody (RVNA) activities ,safety and tolerability of rhRIG vs. HRIG in combination with rabies vaccine for human use (Vero cells) in healthy adult subjects.The study has 7 groups.Subjects will receive rhRIG（20 IU/kg）only, rhRIG（40 IU/kg）only,HRIG（20 IU/kg）only, rhRIG（20 IU/kg）in combination with rabies vaccine for human use, rhRIG（40 IU/kg）in combination with rabies vaccine for human use,HRIG（20 IU/kg）in combination with rabies vaccine for human use,and placebo in combination with rabies vaccine for human use,respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged at least 18 years but not more than 55 years;
2. According to medical history, physical examination and clinical judgment of investigator at enrollment, subjects should have no significant health problems, or their health status or medication treatment remain stable;
3. Subjects and their spouses should use adequate contraceptive methods from the screening day to Day 90;
4. Male subjects must agree not to donate sperm from the first day of enrollment to Day 90;
5. Subjects should sign a written Informed Consent Form;

Exclusion Criteria:

1. Previous exposure or immunization histories of rabies (rabies vaccine and/or immunoglobulin);
2. According to the clinical judgment of investigator, subjects had clinically significant acute disease or infection, including pyrexia (>37.0℃) within 2 weeks before the initial dose;
3. After review of medical history or physical examination results, it is found that subjects have medical histories of abnormalities of heart, liver, kidney, blood, digestive tract, nervous system, spirit and metabolism;
4. Subjects are pregnant or plan to become pregnant or are breast-feeding during the study;
5. According to the judgment of investigator, subjects have clinically significant immunodeficiency or medical history and/or family history of autoimmune disease;
6. According to the judgment of investigator, subjects have known or suspected clinically significant anaphylaxis or hypersensitivity reactions;
7. Immunization has been arranged for the subjects within the next 3 months after the initial dose;
8. Subjects have used immunosuppressive preparations or other immunomodulating agents for more than 14 days within 6 months before the initial dose of study drug;
9. Subjects used hormone agents within 3 days before the initial dose;
10. Subjects donated blood or lost a lot of blood within 56 days before the initial dose;
11. Subjects donated plasma within 7 days before the initial dose;
12. Subjects received transfusion of blood or blood products within 6 months before the initial dose;
13. It is suspected that subjects do not follow study procedures;
14. Intake of alcohol within 12 hours before the initial dose;
15. Subjects smoke more than 20 cigarettes a day;
16. Subjects are obviously allergic to antibiotics;
17. Any other conditions which may affect trial assessment at the discretion of the investigator;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the detection rate of the rabies virus neutralizing antibody (RVNA) activities of rhRIG vs. HRIG in combination with rabies vaccine for human use (Vero cells) in healthy adult subjects | 42 days

SECONDARY OUTCOMES:
Evaluate the rate of adverse reactions of rhRIG or HRIG in combination with rabies vaccine for human use (Vero cells) in healthy subjects | 42 days

REFERENCES:
- [Derived] Li L, Li Y, Bai Y, Li G, Zhang J, Yang L, Zhao W, Zhao W, Luo F, Zhao Q, Zhang Z, Liu Y, Li S, Lu Q, Wang H, Zhang J, Zhang Y, Gao J, Shi N. Neutralizing antibody activity, safety and immunogenicity of human anti-rabies virus monoclonal antibody (Ormutivimab) in Chinese healthy adults: A phase Ⅱb randomized, double-blind, parallel-controlled study. Vaccine. 2022 Oct 6;40(42):6153-6162. doi: 10.1016/j.vaccine.2022.09.022. Epub 2022 Sep 16. PMID 36123259
- [Derived] Zhang J, Shi N, Li G, Li L, Bai Y, Yang L, Zhao W, Gao J, Wei J, Zhao W, Zhai L, Huo P, Ren L, Yu L, Li Y. Population Pharmacodynamic Analyses of Human Anti-Rabies Virus Monoclonal Antibody (Ormutivimab) in Healthy Adult Subjects. Vaccines (Basel). 2022 Jul 29;10(8):1218. doi: 10.3390/vaccines10081218. PMID 36016106